CLINICAL TRIAL: NCT00958308
Title: A Double-blind, Randomized, Placebo-controlled, Single-center Study of the Efficacy and Safety of BIO-K+ CL-1285® in the Prevention of Antibiotic-Associated Diarrhea (AAD) and Clostridium Difficile-Associated Diarrhea (CDAD) in Hospitalized Adult Patients Exposed to Nosocomial Infection
Brief Title: Efficacy and Safety Study in the Prevention of Antibiotic-Associated Diarrhea (AAD) and Clostridium Difficile-Associated Diarrhea (CDAD) in Hospitalized Adult Patients Exposed to Nosocomial Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-SC-9-BIK-01; CL 1285-AAD-CH01
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Antibiotic-Associated Diarrhea; Clostridium Difficile-Associated Diarrhea
Keywords: Probiotic; Antibiotic-Associated Diarrhea (AAD) Prevention; Clostridium Difficile-Associated Diarrhea (CDAD)Prevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Two capsules of placebo (devoid of microorganisms) per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
  Interventions: Other: Placebo
- BIO-K+ CL-1285 (Active Comparator): Two probiotic capsules (BIO-K+ CL-1285®) per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
  Interventions: Other: BIO-K+ CL-1285®
- BIO-K+ CL-1285® & placebo (Other): One probiotic capsule (BIO-K+ CL-1285®) and one placebo capsule (devoid of microorganisms) per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
  Interventions: Other: BIO-K+ CL-1285®; Other: Placebo

INTERVENTIONS:
Other: BIO-K+ CL-1285® — A mixture of Lactobacillus acidophilus and Lactobacillus casei, contains over 50 billion living bacteria per administered dose.
  Arms: BIO-K+ CL-1285; BIO-K+ CL-1285® & placebo
Other: Placebo — Placebo is devoid of microorganisms.
  Arms: BIO-K+ CL-1285® & placebo; Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Bio-K+ CL-1285 in the prevention of Antibiotic-Associated Diarrhea (AAD) and Clostridum difficile-Associated Diarrhea (CDAD) in hospitalized patients exposed to nosocomial infection.

ELIGIBILITY:
Inclusion Criteria:

* Antibiotic therapy for a minimum of 3 days and a maximum of 14 days
* Expected to remain hospitalized for a minimum of 5 days
* Patients who have received less than 36 hours of antibiotic therapy
* Negative pregnancy test at screening
* Obtained his/her informed consent after verbal and written information
* Patients having a telephone available (mobile, work, home)
* Patients having a fridge at home

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients presenting with active diarrhea (3 or more liquid stools per 24 hour period).
* Patients with a history of daily consumption of probiotics, fermented milk and/or yogurt;
* Patients known to have shown a previous reaction, including anaphylaxis, to any substance in composition of the study product (i.e. Non-medicinal ingredients: Cellulose, hypromellose, magnesium stearate (vegetal source), ascorbic acid, Colloidal silicon dioxide)
* Patients presenting with an active, non-controlled intestinal disease such as Crohn's Disease or ulcerative colitis;
* A previous documented C. Difficile infection < 3 months prior to study initiation ;
* Ostomized patients, parenteral nutrition users
* Patients with an immunosuppressive therapy or any health condition causing immunosuppression (including haematological malignancies, acquired immune deficiency syndrome (AIDS))
* Ongoing or recent use of antibiotic therapy in the 30 days prior to the study product first administration.
* Patients with planned administration of antibiotics other than broad spectrum Penicillin, Cephalosporin or Clindamycin for the treatment of an infection;
* Patients with concomitant participation in another clinical trial;
* Patients who are not likely to comply with study requirements

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gao XingWang, MD, Principal Investigator — Xinhua/Yuyao Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

REFERENCES:
- [Result] Gao XW, Mubasher M, Fang CY, Reifer C, Miller LE. Dose-response efficacy of a proprietary probiotic formula of Lactobacillus acidophilus CL1285 and Lactobacillus casei LBC80R for antibiotic-associated diarrhea and Clostridium difficile-associated diarrhea prophylaxis in adult patients. Am J Gastroenterol. 2010 Jul;105(7):1636-41. doi: 10.1038/ajg.2010.11. Epub 2010 Feb 9. PMID 20145608
- See also: Dose-response probiotic study for AAD and CDAD — http://www.ncbi.nlm.nih.gov/pubmed/20145608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1120 patients screened, 255 enrolled at the Xinhua/Yuyao Hospital, Shangai Jiao Tong University, China between Oct. 2008 and March 2009.
Pre-assignment Details: Inclusion & exclusion criterias were used to randomized patients.
Groups:
- BIO-K+ CL-1285® & Placebo: One capsule of probiotic (BIO-K+ CL-1285® with 50 billion colony forming units (CFU)) and one capsule of placebo (devoid of microorganisms) per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
- BIO-K+ CL-1285: Two capsules of probiotic(BIO-K+ CL-1285® - each capsule contains 50 billion CFU) per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
Period: Overall Study
Arm/Group | Placebo | BIO-K+ CL-1285® & Placebo | BIO-K+ CL-1285
Started | 84 | 85 | 86
Completed | 84 | 85 | 86
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BIO-K+ CL-1285® & Placebo | BIO-K+ CL-1285 | Total
Number analyzed (Participants) | 84 | 85 | 86 | 255
Age Continuous [Mean (Standard Deviation); unit: years] | 60.4 (5.88) | 60.2 (6.03) | 60.0 (6.32) | 60 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 40 | 124
  Male | 42 | 43 | 46 | 131
Region of Enrollment [Number; unit: participants]
  China | 84 | 85 | 86 | 255

OUTCOME MEASURES:

1. Primary Outcome: To Assess if Probiotic Prophylaxis (BIO-K+CL1285®) is Effective for the Prevention of AAD in Hospitalized Patients.
Description: Incidence of AAD data were collected using questionnaire and diaries given to participants upon discharge. Diagnosis of AAD was made when a patient produced three or more liquid stools in a 24h period after antibiotic treatment with no other obvious reason for diarrhea.
Time Frame: Up to 40 days
Measure: Number; unit: participants
Groups:
- Placebo: Two capsules of placebo (devoid of microorganisms)per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
- BIO-K+ CL-1285: Two capsules of probiotic (each capsule contains 50 billion CFU) per day. Patients took their daily dose 2h after breakfast and antibiotic administration each day. Patients were then followed for an additionnal 21 days after completion of the assigned intervention.
Arm/Group | Placebo | BIO-K+ CL-1285® & Placebo | BIO-K+ CL-1285
Number analyzed (Participants) | 84 | 85 | 86
participants | 84 | 85 | 86
Statistical Analysis 1: Comparison: Placebo vs BIO-K+ CL-1285® & Placebo vs BIO-K+ CL-1285; The sample size calculation was based on the incidence of AAD. A total of 255 patients was enrolled in order to obtain at least the required 225 evaluable patients.With expected AAD rates of at most 15% - 25% in the treatment groups; and 25% - 35% in the placebo group, these numbers were sufficient to detect the difference in the incidence of AAD between either of the treatment groups vs. placebo with a minimum of 86% statistical power; Test type: Superiority or Other; p = 0.02, Fisher Exact

2. Secondary Outcome: Severity of AAD in Hospitalized Patients Ingesting BIO-K+CL1285® or Placebo.
Description: Duration of diarrhea was determined by number of continuous days of diarrhea. Average number of liquid stools per day was determined by the sum of the number of liquid stools per day in the AAD episode divided by the duration of diarrhea in days.
Time Frame: Up to 40 days
Reporting Status: Not Posted

3. Secondary Outcome: Frequency of Stool Samples Positive for Clostridium Difficile (C. Difficile) Toxin A and/or B.
Description: If diarrhea occured while hospitalized, patients provided a stool sample for C. difficile analysis of Toxin A and/or B. All episodes were recorded by a nurse of clinician on a case report form using the seven-item Bristol Stool Form Scale (Riegler et al., 2001). A diarrhea episode was described as a bowel movement consisting of watery stool with or without solids.
Time Frame: Up to 40 days
Reporting Status: Not Posted

4. Secondary Outcome: Safety Profile of BIO-K+CL1285® Versus Placebo in Hospitalized Patients.
Description: Adverse events were reported by patients in the three study groups.
Time Frame: Up to 40 days
Reporting Status: Not Posted

5. Secondary Outcome: Frequencies of Other Gastrointestinal Symptoms.
Description: Episodes of gastrointestinal disorders during hospitalization were recorded by patient interview and were confirmed by review of patient diaries.
Time Frame: Up to 40 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | BIO-K+ CL-1285® & Placebo | BIO-K+ CL-1285
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/85 | 0/86
Other Adverse Events (participants affected / at risk) | 2/84 | 0/85 | 1/86
OTHER ADVERSE EVENTS (reported when occurring in more than 1.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=84) | BIO-K+ CL-1285® & Placebo (N=85) | BIO-K+ CL-1285 (N=86)
Fever and hematochezia (General disorders) | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less